CLINICAL TRIAL: NCT05409339
Title: Influence of Caffeine Consumption on the Human Circadian System: Neurobehavioral, Hormonal and Cerebral Mechanisms
Brief Title: Influence of Caffeine Consumption on the Human Circadian System
Acronym: CICAFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Carolin Reichert, Principle Investigator, Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CChronobiology
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Caffeine; Caffeine Withdrawal; Sleep; Circadian Rhythm
Keywords: Caffeine; Withdrawal; Sleep; Circadian rhythm
MeSH Terms: interventions — Caffeine; Mannitol

STUDY DESIGN:
Intervention Model Description: The project adopted a double blind, placebo-controlled, randomized within-subjects design. Screenings took place at the Centre for Chronobiology at the Psychiatric University Hospital Basel (UPK, single center). Data collection took place at Clinical Trial Unit, Department of Clinical Research, University of Basel and University Hospital of Basel. Each participant went through three study sessions, i.e. caffeine, placebo, withdrawal. Each of the session consisted of 9 days of pre-ambulatory part, 2 days of laboratory visit, and 7 days of post-ambulatory part.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine-Caffeine (Condition "Caffeine") (Experimental): Through the 9-day pre-ambulatory, 2-day laboratory, and 7-day post-ambulatory parts, participants received 150 mg caffeine x 3 times daily.
  Interventions: Drug: Caffeine
- Caffeine-Placebo (Condition "Withdrawal") (Experimental): During the 9-day ambulatory part, participants received 150 mg caffeine x 3 times daily, followed by a switch to placebo (150 mg mannitol) from the 2nd intake of the 9th day onward, through the laboratory and the post-ambulatory parts.
  Interventions: Drug: Caffeine; Drug: Placebo
- Placebo (Condition "Placebo") (Placebo Comparator): Through the 9-day ambulatory and 2-day laboratory, and 7-day post-ambulatory parts, participants received 150 mg mannitol x 3 times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — 150 mg caffeine, 3 times/day (wakeup + 45 min, +255 min, and +475 min)
  Arms: Caffeine-Caffeine (Condition "Caffeine"); Caffeine-Placebo (Condition "Withdrawal")
Drug: Placebo — Mannitol, 3 times/day (wakeup + 45 min, +255 min, and +475 min)
  Other Names: Mannitol
  Arms: Caffeine-Placebo (Condition "Withdrawal"); Placebo (Condition "Placebo")

SUMMARY:
Surveys indicate that 85% of the adult population consume caffeine on a daily basis. Caffeine acts on sleep homeostatic mechanisms by antagonizing the sleep factor adenosine. Whether and how caffeine also impacts on the circadian regulation of sleep and -wakefulness is fairly unexplored. This study quantifies the influence of regular caffeine intake and its cessation on circadian promotion of sleep and wakefulness, on circadian hormonal markers, well-being, neurobehavioral performance and associated cerebral mechanisms. The knowledge is expected to contribute important insights on recent societal changes in sleep-wake behavior (e.g., shorter sleep duration and delayed sleep phase) and the related increase in people suffering from sleep problems.

DETAILED DESCRIPTION:
Surveys indicate that 85% of the adult population consume caffeine, often on a daily basis. Caffeine acts on sleep homeostatic mechanisms by antagonizing the sleep factor adenosine. Whether and how caffeine also impacts on the circadian regulation of sleep and -wakefulness is fairly unexplored. The circadian timing system promotes wakefulness at the end of the biological day ("wake maintenance zone") and promotes sleep after the onset of the endogenous melatonin secretion ("opening of sleep gate"). There is mounting evidence that circadian and sleep homeostatic mechanisms continuously interact at the neurobehavioral, hormonal and cerebral level. Furthermore, earlier evidence has shown that the strength of circadian wake-promotion and the timing of circadian rhythmicity differs according to a genetic predisposition in the adenosinergic system. Thus, it was assumed that the daily consumption of caffeine may substantially impact on both circadian and homeostatic sleep-wake processes at different systemic levels.

This study aimed at quantifying the influence of regular caffeine intake and its cessation on circadian promotion of sleep and wakefulness, on circadian hormonal markers, well-being, neurobehavioral performance and associated cerebral mechanisms. Specifically, the study investigated the effects of sleep-wake regulatory adaptations to regular caffeine consumption and acute caffeine cessation a) on night-time sleep structure and sleep intensity (electroencephalography, EEG), b) on circadian wake-promotion (nap sleep during the biological day) and circadian timing of hormonal rhythms, and c) on waking quality, as indexed by subjective ratings, objective measures of neurobehavioral performance, and cerebral mechanisms (EEG and functional magnetic resonance imaging [MRI]).

Twenty young healthy regular caffeine consumers were examined in a double-blind, placebo-controlled within-subjects design with three conditions: Regular caffeine intake, regular placebo intake, and cessation of regular caffeine intake. In the laboratory, circadian sleep-wake promotion was assessed by combining EEG and multimodal MRI techniques. Circadian timing was assessed by salivary melatonin and cortisol rhythms. Sleep and waking quality were quantified by continuous polysomnography (during sleep at night and during a nap in the evening), waking EEG, subjective ratings (sleepiness, mood, craving, withdrawal symptoms) and cognitive performance (vigilance and working memory). Each of the three laboratory parts lasted more than 40 h under strictly controlled conditions (i.e., dim light, constant ambient temperature etc.). Subsequent to each laboratory condition, actimetry and sleep diaries served to assess sleep- and waking patterns in the field under caffeine vs. placebo conditions.

The aim was to substantially advance the knowledge about the impact of the commonly encountered caffeine consumption on the sleep-wake regulatory system. Furthermore, the project was intended to substantially contribute to the understanding of complex interplay between sleep-wake regulatory mechanisms in response to acute or long-term changes in the adenosinergic system.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported caffeine consumption: 300 mg - 600 mg daily
* 18-35 years old
* Healthiness

Exclusion criteria based on chronic or debilitating medical conditions:

Normal current health was established based on questionnaires, screenings of urine, and examination by the physician in charge. Given the wide range of illnesses encountered in medical practice, we only list those that were certainly reasons of exclusion:

* Diseases of somatic origin: Cardiovascular-, respiratory-, gastrointestinal-, hematopoietic- visual- and immune system diseases, kidney and urinary tract, endocrine and metabolic diseases, neurologic diseases, infectious diseases, allergies (e.g. skin allergies, acute hay fever), thrombocytopenia or other dysfunction of the blood platelets.
* Sleep disorders: Narcolepsy, sleep apnea (apnea index >10), periodic limb movements (PLMS >15), insomnia (polygraphically recorded sleep efficiency <70 %), hypersomnia, usual time in bed not between 6-9 h (assessed by [101]).
* Chronobiologic disorders: Hypernychthemeral sleep/wake cycle, delayed sleep phase syndrome (waketime >2 h later than desired, or habitually after 10 am), advanced sleep phase syndrome (waketime >2 h earlier than desired or habitually before 5 am).
* Drug/alcohol use, except caffeine: Volunteers must be drug-free (including nicotine and alcohol) for the entire duration of the study, with no history of drug (excluding caffeine) or alcohol dependency.

Exclusion criteria based on to the study requirements:

* Self-reported caffeine consumption: < 300 mg and > 600 mg daily (as estimated from mean caffeine content per serving of caffeine containing beverages and food)
* Body Mass Index (BMI) range: <18 and >26
* Participation in other clinical trials <3 months prior to study begin
* Shift work <3 months prior to study begin
* Transmeridian travel (>2 time zones) <1 month prior to study begin
* Extreme chronotype (Morningness-Eveningness Questionnaire <30 or >70)
* Inability to follow procedures
* Insufficient knowledge of project language (German)

Exclusion criteria based on MRI safety:

* Metallic prosthesis or metallic implants or non-removable objects on the body (e.g. splinters, piercings)
* Tattoos with larger diameter than 10 cm
* Tattoos above the shoulder area
* Claustrophobia
* Contraceptive coil

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Sleep polysomnography in normal baseline sleep | First 8-hour nighttime sleep on the laboratory evening (Day 9)
  Electrophysiological activities were measured by electroencephalography during sleep. Spectral analysis was performed using a Fast-Fourier transformation to quantify delta (0.75 - 4.5 Hz), theta (4.5 - 8 Hz), alpha (8 - 12 Hz), and sigma (12 - 16 Hz), and beta (16 - 32 Hz) power density . Sleep stages, i.e., non-rapid eye-movement (NREM) stage 1, NREM2, NREM3, NREM4, and REM sleep were determined by visual scoring per 30-second epoch in accordance with the guideline of American Academy of Sleep Medicine (AASM).Sleep stages were reported relative to total sleep time. Duration of sleep latencies was also reported.
Sleep polysomnography in an evening nap | approx. 13.5-hour after wake-up time on the laboratory day (Day 10)
  Electrophysiological activities were measured by electroencephalography during the sleep. Spectral analysis was performed using a Fast-Fourier transformation to quantify delta (0.75 - 4.5 Hz), theta (4.5 - 8 Hz), alpha (8 - 12 Hz), and sigma (12 - 16 Hz), and beta (16 - 32 Hz) power density . Sleep stages, i.e., non-rapid eye-movement (NREM) stage 1, NREM2, NREM3, NREM4, and REM sleep were determined by visual scoring per 30-second epoch in accordance with the guideline of American Academy of Sleep Medicine (AASM).Sleep stages were reported relative to total sleep time. Duration of sleep latencies was also reported.
Sleep polysomnography in a recovery sleep | Second 8-hour nighttime sleep following 20-hour wakefulness on the laboratory day (Day 10)
  Electrophysiological activities were measured by electroencephalography during the sleep. A Fast-Fourier Transformation was used to quantify slow wave activities (0.75 - 4.5 Hz), theta (4.5 - 8 Hz), alpha (8 - 12 Hz), and beta (12 - 16 Hz), and sleep stages, i.e., non-rapid eye-movement (NREM) stage 1, NREM2, NREM3, NREM4, and REM sleep were determined by visual scoring through each 30-second epoch in accordance with the guideline of American Academy of Sleep Medicine (AASM).
Wake-EEG | 14 measurements: (Day 9) -130, -20 minutes to the bedtime. (Day 10) +20, +140, +260, +370, +490, +600, +725, +867, +945, +1065, +1180, +1250 minutes after awakening.
  Electrophysiological activities during wakefulness measured by electroencephalography during the sleep. A Fast-Fourier Transformation was used to quantify slow wave activities (0.75 - 4.5 Hz), theta (4.5 - 8 Hz), alpha (8 - 12 Hz), and beta (12 - 16 Hz).
Melatonin levels | 33 samples: (Day 9) -310,-250,-190,-140,-110,-80,-50,-10 minutes to the bedtime. (Day 10) + 50,+110,+170,+230,+290,+350,+400,+460,+515,+580,+610,+670,+700,+735,+765,+935,+965,+995,+1055,+1075,+1115,+1145,+1170, +1190,+1250 after awakening.
  The oscillation of melatonin levels across 43-hour laboratory stay were measured from the 33 salivary samples. The dim-light melatonin onset (DLMO) and average secretion level were analyzed and compared among three conditions.
Subjective sleepiness | 33 samples: (Day 9) -310,-250,-190,-140,-110,-80,-50,-10 minutes to the bedtime. (Day 10) + 50,+110,+170,+230,+290,+350,+400,+460,+515,+580,+610,+670,+700,+735,+765,+935,+965,+995,+1055,+1075,+1115,+1145,+1170, +1190,+1250 after awakening.
  Participants were asked to assess their perceived sleepiness by Karolinska Sleepiness Scale (KSS), where they answered 1 for very alert and 9 for very sleepy.
Vigilance | 7 measurements: (Day 9) -160 minutes to the bedtime. (Day 10) +95, +335, +560, +795, +1040, +1235 minutes after awakening.
  Vigilance was assessed by psychomotor vigilance tasks (PVT). Participants were asked to respond to each stimulus showing on a screen as soon as they can by keying down. The reaction times and lapses were used to indicate the vigilance.
Vigilance-related blood oxygen level-dependent activities | +795 minutes after waking up on the laboratory day (Day 10)
  Regional brain activation is measured by echo-planar-imaging (EPI) sequence in a 3T fMRI scanner during a psychomotor vigilance task (PVT).
Working memory-related blood oxygen level-dependent activities | +775 after waking up on the laboratory day (Day 10)
  Regional brain activation is measured by echo-planar-imaging (EPI) sequence in a 3T fMRI scanner during a working memory task (N-back).
Blood oxygen level-dependent activities in resting state | approx.13.7 hours after waking up on the laboratory day (Day 10)
  Functional connectivity is measured by echo-planar-imaging (EPI) sequence in a 3T fMRI scanner during an eye-open resting state.

SECONDARY OUTCOMES:
Cerebral blood flow | approx. 13.5 hours after waking up on the laboratory day (Day 10)
  Arterial Spin Labeling sequence was used to measure the changes in cerebral blood flow induced by caffeine intake and caffeine cessation.
Caffeine concentrations | 12 samples: (Day 9) -185 minutes to the bedtime. (Day 10) +15, +120, +240, +300, +480, +590, +735, +825, +975, +1085, +1195 minutes after awakening.
  Caffeine concentrations were measured from salivary and perspiratory samples.
Working memory | 7 measurements: (Day 9) -140 minutes to the bedtime. (Day 10) +75, +315, +540, +775, +1020, +1215 minutes after awakening.
  Working memory capacity was measured by N-Back tasks, where participants had a high workload condition (3-back) and a low workload condition (0-back).
Sleep diary | Upon wake-up and bedtime during the ambulatory parts (Day1 to Day8 and Day11 to Day17)
  A daily log was used to record the participant's bed- and wakeup time, self-report sleep quality, tiredness, and activities during the day including caffeine intake.
Actimetry | Constant recording from Day1 to Day17.
  Participants wore an actiwatch to record the muscle tone in order to track the body movement and sleep-wake behaviors constantly throughout the entire study.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Reichert, Dr., Principal Investigator — UPK Basel
Locations (1):
- UPK Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Weibel J, Lin YS, Landolt HP, Garbazza C, Kolodyazhniy V, Kistler J, Rehm S, Rentsch K, Borgwardt S, Cajochen C, Reichert CF. Caffeine-dependent changes of sleep-wake regulation: Evidence for adaptation after repeated intake. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109851. doi: 10.1016/j.pnpbp.2019.109851. Epub 2019 Dec 19. PMID 31866308
- [Result] Weibel J, Lin YS, Landolt HP, Kistler J, Rehm S, Rentsch KM, Slawik H, Borgwardt S, Cajochen C, Reichert CF. The impact of daily caffeine intake on nighttime sleep in young adult men. Sci Rep. 2021 Feb 25;11(1):4668. doi: 10.1038/s41598-021-84088-x. PMID 33633278
- [Result] Weibel J, Lin YS, Landolt HP, Berthomier C, Brandewinder M, Kistler J, Rehm S, Rentsch KM, Meyer M, Borgwardt S, Cajochen C, Reichert CF. Regular Caffeine Intake Delays REM Sleep Promotion and Attenuates Sleep Quality in Healthy Men. J Biol Rhythms. 2021 Aug;36(4):384-394. doi: 10.1177/07487304211013995. Epub 2021 May 23. PMID 34024173
- [Result] Lin YS, Weibel J, Landolt HP, Santini F, Garbazza C, Kistler J, Rehm S, Rentsch K, Borgwardt S, Cajochen C, Reichert CF. Time to Recover From Daily Caffeine Intake. Front Nutr. 2022 Feb 2;8:787225. doi: 10.3389/fnut.2021.787225. eCollection 2021. PMID 35187019
- [Result] Lin YS, Weibel J, Landolt HP, Santini F, Meyer M, Brunmair J, Meier-Menches SM, Gerner C, Borgwardt S, Cajochen C, Reichert C. Daily Caffeine Intake Induces Concentration-Dependent Medial Temporal Plasticity in Humans: A Multimodal Double-Blind Randomized Controlled Trial. Cereb Cortex. 2021 May 10;31(6):3096-3106. doi: 10.1093/cercor/bhab005. PMID 33585896